CLINICAL TRIAL: NCT03992131
Title: SEASTAR: A Phase 1b/2, Open-label, Parallel Arm Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Oral Rucaparib in Combination With Other Anticancer Agents in Patients With a Solid Tumor
Brief Title: A Study to Evaluate Rucaparib in Combination With Other Anticancer Agents in Participants With a Solid Tumor (SEASTAR)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to a change in development priorities, no further clinical development of the lucitanib plus rucaparib or lucitanib plus sacituzumab govitecan combinations is planned at this time.
Sponsor: pharmaand GmbH (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-098; 2018-003759-39 (EudraCT Number)
Record Dates: First submitted 2019-06-04; First posted 2019-06-20 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Triple-negative Breast Cancer; Urothelial Carcinoma; Solid Tumor
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell | interventions — rucaparib; E-3810; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Rucaparib and Lucitanib (Experimental): Participants will receive oral rucaparib twice daily (BID) and oral lucitanib once daily (QD) continuously in 28-day cycles.
  Interventions: Drug: Rucaparib; Drug: Lucitanib
- Arm B: Rucaparib BID and Sacituzumab Govitecan (Experimental): Participants will receive oral rucaparib BID, administered continuously, in combination with intravenous (IV) sacituzumab govitecan administration on Day 1 and Day 8 of a 21-day cycle.
  Interventions: Drug: Rucaparib; Drug: Sacituzumab govitecan
- Arm B: Rucaparib QD and Sacituzumab Govitecan (Experimental): Participants will receive oral rucaparib QD, administered continuously, in combination with IV sacituzumab govitecan administration on Day 1 and Day 8 of a 21-day cycle.
  Interventions: Drug: Rucaparib; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Rucaparib — Rucaparib will be administered per schedule specified in the arm description.
  Other Names: Rubraca; CO-338
Drug: Lucitanib — Lucitanib will be administered per schedule specified in the arm description.
  Other Names: CO-3810
  Arms: Arm A: Rucaparib and Lucitanib
Drug: Sacituzumab govitecan — Sacituzumab govitecan will be administered per schedule specified in the arm description.
  Other Names: IMMU-132
  Arms: Arm B: Rucaparib BID and Sacituzumab Govitecan; Arm B: Rucaparib QD and Sacituzumab Govitecan

SUMMARY:
This is an open label, Phase 1b/2 study with multiple treatment arms evaluating the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of rucaparib in combination with a second anticancer therapy in participants with an advanced/metastatic solid malignancy (Phase 1b), followed by evaluation of the combination in one or more specific participant populations in an expansion phase (Phase 2 cohorts).

ELIGIBILITY:
Inclusion Criteria Phase 1b (all arms):

* Solid tumor, advanced or metastatic, progressed on standard treatment participants in Arm B must have either triple negative breast cancer OR urothelial carcinoma OR ovarian cancer OR have a solid tumor with a deleterious mutation in BRCA1, BRCA2, PALB2, RAD51C or RAD51D
* Measurable disease per RECIST v1.1
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Tumor tissue for genomic analysis

Exclusion Criteria Phase 1b (all arms):

* Known history of myelodysplastic syndrome (MDS)
* Symptomatic and/or untreated central nervous system (CNS) metastases

Inclusion Criteria Phase 2 (all arms):

* Histologically or cytologically confirmed solid tumor, previously treated and measurable per RECIST v1.1, as follows:
* Arm A: ovarian cancer with gBRCAwt disease, either platinum-sensitive OR platinum-resistant
* Arm B: Metastatic triple negative breast cancer OR advanced/ metastatic urothelial carcinoma OR relapsed ovarian cancer
* At least 1 prior line of standard therapy for advanced disease
* Adequate organ function
* ECOG 0 or 1
* Tumor tissue for genomic analysis

Exclusion Criteria Phase 2 (all arms):

* Prior poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor treatment allowed for participants with ovarian cancer
* Known history of MDS
* Symptomatic and/or untreated CNS metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 phases: Phase 1b and Phase 2. Enrollment was terminated before Phase 1b was complete, due to Sponsor's decision to discontinue development of the combination of rucaparib and sacituzumab govitecan. Hence, Phase 2 portion of the study was not conducted.
Groups:
- Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD: Participants received oral rucaparib 300 milligrams (mg) twice daily (BID) and oral lucitanib 4 mg once daily (QD) continuously in 28-day cycles.
- Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD: Participants received oral rucaparib 400 mg BID and oral lucitanib 4 mg QD continuously in 28-day cycles.
- Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD: Participants received oral rucaparib 400 mg BID and oral lucitanib 6 mg QD continuously in 28-day cycles.
- Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD: Participants received oral rucaparib 600 mg BID and oral lucitanib 6 mg QD continuously in 28-day cycles.
- Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan: Participants received oral rucaparib 300 mg BID, administered continuously, in combination with intravenous (IV) sacituzumab govitecan 6 mg/kilogram (kg) administration on Day 1 and Day 8 of a 21-day cycle.
- Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan: Participants received oral rucaparib 300 mg QD, administered continuously, in combination with IV sacituzumab govitecan 6 mg/kg administration on Day 1 and Day 8 of a 21-day cycle.
Period: Overall Study
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan
Started | 6 | 4 | 3 | 6 | 3 | 3
Received at Least 1 Dose of Study Drug | 6 | 4 | 3 | 6 | 3 | 3
Completed | 6 | 4 | 3 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who have received at least 1 dose of study drug.
Groups:
- Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD: Participants received oral rucaparib 300 mg BID and oral lucitanib 4 mg QD continuously in 28-day cycles.
- Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan: Participants received oral rucaparib 300 mg BID, administered continuously, in combination with IV sacituzumab govitecan 6 mg/kg administration on Day 1 and Day 8 of a 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan | Total
Number analyzed (Participants) | 6 | 4 | 3 | 6 | 3 | 3 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 0 | 6 | 3 | 2 | 17
  >=65 years | 3 | 1 | 3 | 0 | 0 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 5 | 2 | 3 | 19
  Male | 1 | 2 | 1 | 1 | 1 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 5 | 4 | 2 | 4 | 3 | 3 | 21
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 0 | 0 | 3
  White | 5 | 3 | 2 | 4 | 2 | 3 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response, as Assessed by the Investigator Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1 (Phase 2)
Description: Objective response was defined as a documented and confirmed best overall response of complete response (CR) or partial response (PR) as assessed by the investigator. CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 millimeters (mm); and normalization of tumor marker level. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: From the first dose of study drug until the date of documented response to treatment, assessed up to 2 years
Population: Due to Sponsor's decision to discontinue development of the combination of rucaparib and sacituzumab govitecan, the study was terminated before Phase 1b was complete, and Phase 2 portion of the study was not conducted. Hence, the data for this outcome measure could not be collected and analyzed.
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Duration of Response (DOR) (Phase 2)
Description: Duration of response was measured from the date that best response (CR or PR) was first recorded until the first date that disease progression was documented per RECIST v1.1. CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm; and normalization of tumor marker level. PR: At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD. Progressive disease: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions was also considered progression.
Time Frame: From the date of first best response to disease progression or death, whichever occurs first, assessed up to 2 years
Population: as for outcome 1
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Progression-free Survival (PFS) (Phase 2)
Description: PFS was measured as the 1+ the number of days from the first dose of study drug to documented radiographic progression, according to RECIST v1.1, as determined by the investigator, or death due to any cause, whichever occurred first. Progressive disease: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions was also considered progression.
Time Frame: From the first dose of study drug to documented radiographic progression or death, whichever occurs first, assessed up to 2 years
Population: as for outcome 1
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Objective Response, as Assessed by the Investigator Per RECIST v1.1 (Phase 1b)
Description: Objective response was defined as a documented and confirmed best overall response of CR or PR as assessed by the investigator. CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm; and normalization of tumor marker level. PR: At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: From the first dose of study drug until the date of documented response to treatment, assessed up to 2 years
Population: Efficacy population included all participants who had received at least 1 dose of rucaparib or the second study drug and who had measurable disease per RECIST v1.1 at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan
Number analyzed (Participants) | 6 | 4 | 3 | 6 | 3 | 3
Participants | 1 | 0 | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 2 years
Description: Safety population included all participants who have received at least 1 dose of study drug.
Arm/Group | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/3 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/4 | 0/3 | 2/6 | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 3/3 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD (N=6) | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD (N=4) | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD (N=3) | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD (N=6) | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan (N=3) | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Rucaparib 300 mg BID and Lucitanib 4 mg QD (N=6) | Arm A2: Rucaparib 400 mg BID and Lucitanib 4 mg QD (N=4) | Arm A3: Rucaparib 400 mg BID and Lucitanib 6 mg QD (N=3) | Arm A4: Rucaparib 600 mg BID and Lucitanib 6 mg QD (N=6) | Arm B1: Rucaparib 300 mg BID and Sacituzumab Govitecan (N=3) | Arm B2: Rucaparib 300 mg QD and Sacituzumab Govitecan (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 3 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 2 | 2
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 1 | 2 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 1 | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 2 | 1 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 2 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0 | 1 | 2 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 2 | 2 | 4 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to Sponsor's decision to discontinue development of the combination of rucaparib and sacituzumab govitecan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03992131/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT03992131/SAP_001.pdf